CLINICAL TRIAL: NCT06949410
Title: Phase I Trial of a Chimeric (Trastuzumab-like and Pertuzumab-like) HER2 B Cell Peptide Vaccine Emulsified in ISA 720 Adjuvant for Locally Advanced HER2 Positive Breast Cancer
Brief Title: HER2 Vaccine for Locally Advanced Breast Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pravin T.P Kaumaya (Other)
Responsible Party: Sponsor-Investigator, Pravin T.P Kaumaya, The Vera Bradley Foundation Endowed Chair in Breast Cancer Innovation Professor of Microbiology & Immunology, Indiana University
Organization: Indiana University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTO-IUSCCC-0864
Record Dates: First submitted 2025-04-22; First posted 2025-04-29 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer; HER2-positive Breast Cancer
Keywords: vaccine; immune system; immunotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — CHP-HER2 vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- HER2 Vaccine Arm (Experimental): MVF-HER2 266-296 and MVF HER2 597-626 peptide vaccines are combined in 1.5 mg doses of each peptide into a 3.0 mg total dose. This is administered intramuscularly in the gluteus maximus once every 21 days for three doses, in alternating sides (i.e. left->right->left), with a booster administered at 6 months.
  Interventions: Drug: HER2 Vaccine

INTERVENTIONS:
Drug: HER2 Vaccine — MVF-HER2 266-296 and MVF HER2 597-626 peptide vaccines

SUMMARY:
The goal of this study is to test an investigational vaccine to activate the immune system to fight breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years old at the time of informed consent
2. Ability to provide written informed consent and HIPAA authorization CTO-IUSCC-0864
3. Histologically confirmed HER2 positive breast cancer

   1. Any Estrogen Receptor/Progesterone Receptor status is allowed.
   2. HER2 positive is defined as HER2 3+ by immunohistochemistry (IHC) or 2+ by IHC associated with a fluorescence in situ hybridization (FISH) ratio of > 2.0 or > 6 total HER2 gene copies per cell.
4. High-risk disease defined as one of the following:

   1. Any residual invasive carcinoma in the breast or axillary nodes in the final pathology from resected tumor following neoadjuvant taxane and trastuzumab-based chemotherapy
   2. Inflammatory phenotype at the time of diagnosis per the treating physician
   3. Clinical stage III disease at the time of diagnosis per the treating physician and/or clinical imaging
   4. Locally recurrent disease and have undergone definitive local therapy
5. Received at least six months of HER2 targeted therapy with trastuzmab +/- pertuzumab TDM-1, or others in the neoadjuvant or adjuvant setting

   a. Any combination of HER2 targeted therapy in the curative setting is allowed, including neratinib or others on a clinical trial
6. Completed last dose of HER2 targeted therapy no more than 6 months prior to registration
7. Completed last dose of cytotoxic chemotherapy or radiation at least 30 days prior to registration with resolution of any prior toxicity to ≤ 2 with the exception of alopecia
8. ECOG performance status of 0 to 2
9. Adequate organ function as indicated by:

   1. Total bilirubin < 1.5 mg/dL (except in patients with documented Gilbert's disease, who must have a total bilirubin < 3.0 mg/dL)
   2. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2.0 x ULN
   3. Calculated creatinine clearance of > 60 mL/min using the Cockcroft-Gault formula
   4. Absolute neutrophil count (ANC) > 1.0 K/mm3
   5. Platelets > 100 K/ mm3
10. Adequate cardiac function defined as left ventricular ejection fraction (LVEF) above the institutional lower limit of normal by echocardiogram or MUGA obtained within 90 days of registration
11. Women of childbearing potential must have a negative serum pregnancy test within 14 days of protocol registration. Women are considered to have childbearing potential (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) unless they meet one of the following criteria:

    1. Has undergone a hysterectomy or bilateral oophorectomy; or
    2. Has been naturally amenorrheic for at least 12 consecutive months.
12. Women of childbearing potential and men must agree to use one effective contraception throughout the study and for 6 months after the last study treatment.

Note: Acceptable methods of birth control include abstinence, partner with previous vasectomy, placement of an intrauterine device (IUD), condom with spermicidal foam/gel/film/cream/suppository, diaphragm or cervical vault cap, or hormonal birth control (pills or injections).

Exclusion Criteria:

1. Any distant disease recurrence.
2. Patients with active malignancy other than breast cancer. Note: Patients with prior malignancies without recurrence after standard treatment will not be excluded.
3. Patients receiving or planned to receive adjuvant CDK4/6 inhibitor therapy
4. Patients who are {MVF-HER-2(266-296) and MVF-HER-2 (597-626)} immediate hypersensitivity skin test positive.
5. Patients who require or likely to require corticosteroids or other immunosuppressives
6. Patients with active autoimmune diseases including rheumatoid arthritis, systemic lupus erythematosus, scleroderma, polymyositis dermato-myositis, or a vasculitic syndrome.

   Note: At the discretion of the treating physician, patients who show disease control for at least 6 months and do not require immunosuppressives may be enrolled.
7. Patients who have developed anaphylactic responses to other vaccines.
8. Patients who have evidence of active infection that requires antibiotic therapy. Patients must have been off antibiotic treatment for at least 3 weeks prior to initiating treatment and must be confirmed to be clear of the infection.
9. Known seropositive or active viral infection with human immunodeficiency virus (HIV), hepatitis B (HBV), or hepatitis C (HCV). Seropositivity due to vaccination are eligible.
10. Uncontrolled illness that would limit safety or compliance with study procedures including, but not limited to, active infection, congestive heart failure, unstable angina, or cardiac arrhythmia.
11. Patients with serious uncontrolled cardiopulmonary disorders, including congestive heart failure, symptomatic coronary artery disease, serious cardiac arrhythmia, and symptomatic chronic obstructive pulmonary disease or patients with other serious uncontrolled medical diseases. At the discretion of the treating physician, patients who show disease control for at least 6 months may be enrolled.
12. History of splenectomy
13. Pregnant or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2029-12 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Evaluation of safety and toxicity at regular intervals by NCI common toxicity criteria 5.0 | through completion of 3 vaccine series (i.e. up to day 64 post final vaccine injection)
  Number of adverse events as assessed by the NCI CTCAE v. 5.0
Immune Response | through completion of 3 vaccine series (i.e. up to day 64 post final vaccine injection)
  Humoral immune response will be measured by ELISA quantification of IgM and IgG antibodies to HER2 (597-626) and HER2 (266-296).

CONTACTS AND LOCATIONS:
Overall Officials: Pravin Kaumaya, PhD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Melvin & Bren Simon Comprehensive Cancer Center, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided